CLINICAL TRIAL: NCT01259674
Title: Randomized, Single-center, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Tolerability of ABO/MEG-B-09 in Pediatric Cough
Brief Title: Evaluation of the Efficacy and Tolerability of ABO/MEG-B-09 in Children With Acute Cough
Acronym: ABOMEG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB-Resp-09
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Cough
Keywords: Pediatric; children; acute cough; treatment; syrup; protective natural extracts
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AboMeg-B-09 syrup (Experimental): Syrup: AboMeg-B-09 5ml to be taken 4 times a day during the entire study period
  Interventions: Device: AboMeg-B-09
- Placebo (Placebo Comparator): Placebo syrup
  Interventions: Other: Placebo

INTERVENTIONS:
Device: AboMeg-B-09 — Syrup: AboMeg-B-09 5ml to be taken 4 times a day during the entire study period
  Arms: AboMeg-B-09 syrup
Other: Placebo — Placebo syrup: 5ml to be taken 4 times a day during the entire study period
  Arms: Placebo

SUMMARY:
The present clinical trial will examine the use of ABO/MEG-B-09 syrup in children with acute cough as compared to a placebo syrup.

DETAILED DESCRIPTION:
Subjects will be asked to take 4 doses of 5 ml containing a mixture of honey and other natural ingredients or a placebo syrup everyday, during 8 days. The following outcomes will be noted down in a diary: occurence and severity of diurnal and nocturnal cough events (cough score) and symptoms, impediment of normal life activities (school, sleeping), the number of medical visits and type of medication needed if any.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 and 6
* Acute cough - lasting 1-3 weeks
* Written informed consent by the parents/legal tutors
* Parents/legal tutors must be willing not to give to the child other medications or products for the treatment of cough during the study period, unless they become clinically indicated in which case a rescue regimen can be administered and the child will be withdrawn from the study
* Parents/legal tutors must be willing to comply with the study protocol

Exclusion Criteria:

* Children treated with immunostimulators and immune regulating drugs during the last month before starting the study
* Children with immunodeficiencies or immune suppression
* Children with chronic diseases - Pulmonary Diseases, Renal insufficiency, Heart diseases
* Children treated with antibiotics, including prophylactic treatment
* Children being treated with systemic corticosteroids - including oral aerosol inhaler
* Children with potential immunosuppressive viral diseases - Measles, Chickenpox, Rubella, Infectious mononucleosis - within the last month
* Children who have participated in previous studies with experimental products within the last month
* Children with asthma or suspected diagnosis of asthma
* Children with bacterial diseases - Pneumonia, Sepsis
* Children with diabetes because of the high content of sugar of the study products - ABO/MEG-B-09 and placebo
* Children allergic to any study product ingredients
* Children/Parents/legal tutors with psychological condition that may, in the investigator's opinion, adversely affect their co-operation with the study protocol - syrup administration or compilation of the diary

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Cough score variation | Measured at Baseline Visit (day 0) and at the Last Visit (day 8)
  Clinical diurnal and nocturnal cough score (Chung)

SECONDARY OUTCOMES:
Cough reflex sensitivity | Measured at Baseline Visit (day 0) and at the Last Visit (day 8)
  Capsaicin test - Cough Reflex Index (CRI) -
Objective breath sounds | Measured at Baseline Visit (day 0) and at the Last Visit (day 8)
  Wheezometer test
The ventilation of the various pulmonary zones | Measured at Baseline Visit (day 0) and at the Last Visit (day 8)
  Vibration Response Imaging (VRI) xp test
Quality of life | Measured at Baseline Visit (day 0) and at the Last Visit (day 8)
  Quality of life questionnaire (QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Arienne de Jong, PhD, Study Chair — Sprim Advanced Life Sciences
Locations (1):
- Santa Maria della Misercordia di Udine Hospital, Udine, Udine, Italy